CLINICAL TRIAL: NCT07153861
Title: Oral Mucosal Graft Versus Labial Graft in Female Urethroplasty: A Prospective Comparative Study
Brief Title: Oral Mucosal Graft Versus Labial Graft in Female Urethroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Ahmed Elmaadawy, Lecturer of Urology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR1113/2/25
Record Dates: First submitted 2025-08-24; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Oral Mucosal Graft; Labial Graft; Female; Urethroplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Patients will be admitted for the surgical management by the oral mucosal graft urethroplasty with the anterior onlay technique.
  Interventions: Procedure: Oral mucosal graft
- Group 2 (Experimental): Patients will be admitted for the surgical management by the labial graft urethroplasty with the anterior onlay technique.
  Interventions: Procedure: Labial graft

INTERVENTIONS:
Procedure: Oral mucosal graft — Patients will be admitted for the surgical management by the oral mucosal graft urethroplasty with the anterior onlay technique.
  Arms: Group 1
Procedure: Labial graft — Patients will be admitted for the surgical management by the labial graft urethroplasty with the anterior onlay technique.
  Arms: Group 2

SUMMARY:
This study aims to compare the oral versus labial graft in female urethroplasty in female urethral stricture.

DETAILED DESCRIPTION:
Female urethral stricture is an uncommon condition with an estimated prevalence of 4%-13% in women with bladder outlet obstruction.

Urethral reconstruction may become the treatment of choice in stricture recurrence following the failure of minimally invasive procedures. and the use of flaps and grafts has all been proposed. Different materials (e.g., vaginal and genital mucosal graft or flap, bladder mucosal flap, and oral mucosal graft) have been reported for augmentation urethroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with urethral stricture.
* Female patients with non-traumatic urethral stricture.

Exclusion Criteria:

* Female patients with traumatic urethral stricture.
* Female patients with systemic contraindications of surgery like bleeding disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female undergoing urethroplasty
Enrollment: 40 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Urine flow rate | 6 months post-procedure
  Urine flow rate will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.